CLINICAL TRIAL: NCT05795803
Title: Effects of a Pandemic Forced Isolation Context on Adolescents With Somatic Symptom Disorder. A Panel Study
Brief Title: Effects of COVID-19 Forced Isolation Context on Adolescents With and Without Somatic Symptom Disorder
Status: Completed | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 11/2020
Record Dates: First submitted 2020-05-11; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Somatic Symptom Disorder
Keywords: SSD; adolescents; coping strategies; social media

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SSD group: Adolescents with SSD diagnosis made within previously six months or before unless assessed and confirmed by a specialist within the last six months
  Interventions: Other: Forced isolation context
- Without SSD group: Control group: adolescents without diagnosis of SSD, matched with the SSD group by age and sex
  Interventions: Other: Forced isolation context

INTERVENTIONS:
Other: Forced isolation context — Exposure to the forced isolation context provided by the ongoing Covid-19 pandemic restrictive measures
  Other Names: COVID-19 lockdown

SUMMARY:
The purpose of this study is to evaluate whether a forced isolation context (such provided by the ongoing Covid-19 pandemic restrictive measures) could reduce the burden of somatic symptoms among a group of patients with Somatic Symptom Disorder (SSD). Secondary objective is to assess if a reduction in terms of depression tendency and anxiety occurs in this specific population and which are the effect of such a context among a group of adolescents without SSD. We want to compare these results with data obtained at the end of the pandemic.

DETAILED DESCRIPTION:
This study aims to evaluate whether the forced isolation context provided by the ongoing Covid-19 pandemic is providing an advantage in terms of reduction of somatic symptoms burden among an Italian group of adolescents with SSD, assessed by the Patient Health Questionnaire (PhQ15) administered during and at the end of the pandemic.

Secondary objectives of the study are:

* To investigate the difference in anxiety and depression scores assessed by the Multidimensional Anxiety Scale for Children (MASC2) and Child Development Inventory (CDI-2) questionnaires among a group of SSD adolescents, during and after the pandemic isolation context.
* To investigate the difference in anxiety and depression scores assessed by the Multidimensional Anxiety Scale for Children (MASC2) and Child Development Inventory (CDI-2) questionnaires among a group of adolescents without SSD, during and after the pandemic isolation context.
* To compare the difference in anxiety and depression scores time modification between the two groups of adolescents.
* To explore through tailored questions which adolescents' coping strategies are during a pandemic isolation context among SSD patients and a group of controls without SSD.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged between 12 and 17 years old who received a diagnosis of SSD within the last six months or before unless assessed and confirmed by a specialist within the last six months
* Adolescents without a diagnosis of SSD, who previously accessed the Institute for maternal and child health "Burlo Garofolo" Emergency Department for traumatic injuries or the Pediatric Clinic/Day Hospital Service for oral immunotherapy because of food allergies.
* Adolescents experiencing a quarantine period during the Covid19 pandemic.

Exclusion Criteria:

* Adolescents with cognitive impairment.
* Adolescents with chronic diseases.
* Adolescents with other neuropsychiatric disorders according to the fifth edition of the Diagnostic and Statistical Manual of Mental Disorder (DSM V).
* For the group without SSD diagnosis, any access to Emergency Department for unexplained chronic pain or any history of other psychiatric comorbidities.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: * SSD group: Adolescents who received a diagnosis of SSD at the Institute for maternal and child health "Burlo Garofolo"
  * Without SSD group: Adolescents who accessed the Emergency Department for traumatic injuries or the Pediatric Clinic/Day Hospital Service for oral immunotherapy because of food allergies.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Difference in mean PhQ15 scale scores between T0 and T1 in the SSD adolescents group. | During the pandemic and within 6 months after the end
  To SSD group, the Health Questionnaire Physical Symptoms (PhQ15) will be administrated to quantify the somatic symptom burden.

SECONDARY OUTCOMES:
Difference in mean MASC2 scores between T0 and T1 in the SSD group. | During the pandemic and within 6 months after the end
  SSD adolescents will receive the Multidimensional Anxiety Scale for Children (MASC 2), composed by 50 items, to quantify adolescents' anxiety.
Difference in mean CDI-2 short questionnaire scores between T0 and T1 in the SSD group. | During the pandemic and within 6 months after the end
  SSD adolescents will receive the Children's Depression Inventory (CDI-2) self-report short questionnaire, composed by 12 items, to quantify adolescents' depression.
Difference in mean MASC2 scores between T0 and T1 in the adolescents group without SSD diagnosis. | During the pandemic and within 6 months after the end
  Adolescents without SSD will receive the Multidimensional Anxiety Scale for Children (MASC 2), composed by 50 items, to quantify adolescents' anxiety
Difference in mean CDI-2 short questionnaires scores between T0 and T1 in the adolescents group without SSD diagnosis. | During the pandemic and within 6 months after the end
  Adolescents without SSD will receive the Children's Depression Inventory (CDI-2) self-report short questionnaire, composed by 12 items, to quantify adolescents' depression
Comparison between the two groups of adolescents in the mean T1-T0 differences for MASC2 scores. | During the pandemic and within 6 months after the end
  Differences in the Multidimensional Anxiety Scale for Children (MASC 2), composed by 50 items
Comparison between the two groups of adolescents in the mean T1-T0 differences for CDI-2 short questionnaires scores. | During the pandemic and within 6 months after the end
  Differences in Children's Depression Inventory (CDI-2) self-report short questionnaire, composed by 12 items
Description of adolescents' coping strategies during a pandemic isolation context among SSD and non-SSD adolescent | During the pandemic
  A general anonymous semi-structured survey will be administered to both the groups in order to investigate their habits, social media and videogames pattern of usage, and other leisure pattern of frequency. This will provide us a description of adolescents' general coping strategies during quarantine period.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Abbracciavento, MD, Study Chair — Institute for maternal and child health Burlo Garofolo; Laura De Nardi, MD, Principal Investigator — Institute for maternal and child health Burlo Garofolo; Andrea Trombetta, MD, Principal Investigator — Institute for maternal and child health Burlo Garofolo
Locations (1):
- Institute for Maternal and Child Health - IRCCS Burlo Garofolo-, Trieste, Italy